CLINICAL TRIAL: NCT04198948
Title: Interaction Between Omeprazole and Gliclazide in CYP2C19 Normal/ Ultrarapid Metabolisers
Acronym: INTERGLIKOM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sarajevo (Other)
Collaborators: General Hospital Prim. Dr. Abdulah Nakas (Other); University of Dundee (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Tanja Dujic, PhD, Associate Professor, University of Sarajevo
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 0101-3678/18; 209943/Z/17/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Results first posted 2021-07-15 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Omeprazole; Gliclazide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole, Then Placebo (Experimental): Healthy volunteers, CYP2C19 extensive/ultrarapid metabolisers, will receive 20 mg of omeprazole alone for 4 days, and concomitantly with single dose of gliclazide on day 5. After a wash-out period, they will receive placebo under same conditions in a cross-over manner.
  Interventions: Drug: Omeprazole; Drug: Placebo oral tablet; Drug: Gliclazide
- Placebo, Then Omeprazole (Experimental): Healthy volunteers, CYP2C19 extensive/ultrarapid metabolisers, will receive placebo alone for 4 days, and concomitantly with single dose of gliclazide on day 5. After a wash-out period, they will receive omeprazole under same conditions in a cross-over manner.
  Interventions: Drug: Omeprazole; Drug: Placebo oral tablet; Drug: Gliclazide

INTERVENTIONS:
Drug: Omeprazole — Omeprazole (20 mg) will be administered orally once daily for 5 days in one of the two treatment periods.
Drug: Placebo oral tablet — Placebo will be administered orally once daily for 5 days in one of the two treatment periods.
Drug: Gliclazide — Gliclazide (40 mg) will be administered orally once, concomitantly with omeprazole or placebo on day 5.

SUMMARY:
Proton pump inhibitors (PPIs) are treatment of choice for different gastrointestinal disorders common in type 2 diabetes. Sulfonylureas (SUs) are anti-diabetes agents particularly widely used in developing countries. Gliclazide, a recommended SU drug, is metabolised in part by CYP2C19, the main enzyme responsible for the PPI metabolism.

A randomised, placebo-controlled, two-sequence, two-period crossover study will be performed to explore whether gliclazide pharmacokinetics (PK) and pharmacodynamics (PD) are altered upon co-administration with omeprazole. Sixteen healthy volunteers, CYP2C19 extensive/ultrarapid metabolisers (EM/UM), will receive placebo or omeprazole alone for 4 days, and concomitantly with single dose of gliclazide on day 5. Plasma concentration of gliclazide will be measured for 24 hours, and plasma glucose and insulin levels up to 12 hours after gliclazide administration.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Age 18-30 years
* Non-smokers
* CYP2C19 extensive/ultrarapid metabolisers

Exclusion Criteria:

* medical history of hepatic, renal, gastrointestinal and hematologic disease or any acute or chronic disease, or drug allergy to sulfonylureas or PPIs or history of drug abuse
* abnormalities in physical examination, ECG and routine clinical laboratory tests (including fasting blood glucose concentration)
* medication use during the 14 days prior and during the study period
* grapefruit, grapefruit juice, alcohol, beverages or food containing methylxanthines use during 72 h prior and during the study period

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Dujic, PhD, Principal Investigator — University of Sarajevo; Aida Kulo Cesic, PhD, Principal Investigator — University of Sarajevo
Locations (1):
- General Hospital Prim. Dr. Abdulah Nakas, Sarajevo, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Kalra S, Aamir AH, Raza A, Das AK, Azad Khan AK, Shrestha D, Qureshi MF, Md Fariduddin, Pathan MF, Jawad F, Bhattarai J, Tandon N, Somasundaram N, Katulanda P, Sahay R, Dhungel S, Bajaj S, Chowdhury S, Ghosh S, Madhu SV, Ahmed T, Bulughapitiya U. Place of sulfonylureas in the management of type 2 diabetes mellitus in South Asia: A consensus statement. Indian J Endocrinol Metab. 2015 Sep-Oct;19(5):577-96. doi: 10.4103/2230-8210.163171. PMID 26425465
- [Background] Schopman JE, Simon AC, Hoefnagel SJ, Hoekstra JB, Scholten RJ, Holleman F. The incidence of mild and severe hypoglycaemia in patients with type 2 diabetes mellitus treated with sulfonylureas: a systematic review and meta-analysis. Diabetes Metab Res Rev. 2014 Jan;30(1):11-22. doi: 10.1002/dmrr.2470. PMID 24030920
- [Background] Zhang Y, Si D, Chen X, Lin N, Guo Y, Zhou H, Zhong D. Influence of CYP2C9 and CYP2C19 genetic polymorphisms on pharmacokinetics of gliclazide MR in Chinese subjects. Br J Clin Pharmacol. 2007 Jul;64(1):67-74. doi: 10.1111/j.1365-2125.2007.02846.x. Epub 2007 Feb 12. PMID 17298483
- [Background] Shao H, Ren XM, Liu NF, Chen GM, Li WL, Zhai ZH, Wang DW. Influence of CYP2C9 and CYP2C19 genetic polymorphisms on pharmacokinetics and pharmacodynamics of gliclazide in healthy Chinese Han volunteers. J Clin Pharm Ther. 2010 Jun;35(3):351-60. doi: 10.1111/j.1365-2710.2009.01134.x. PMID 20831536
- [Background] Sun XM, Tan JC, Zhu Y, Lin L. Association between diabetes mellitus and gastroesophageal reflux disease: A meta-analysis. World J Gastroenterol. 2015 Mar 14;21(10):3085-92. doi: 10.3748/wjg.v21.i10.3085. PMID 25780309
- [Background] Furuta T, Iwaki T, Umemura K. Influences of different proton pump inhibitors on the anti-platelet function of clopidogrel in relation to CYP2C19 genotypes. Br J Clin Pharmacol. 2010 Sep;70(3):383-92. doi: 10.1111/j.1365-2125.2010.03717.x. PMID 20716239
- [Background] Dujic T, Zhou K, Donnelly LA, Leese G, Palmer CNA, Pearson ER. Interaction between variants in the CYP2C9 and POR genes and the risk of sulfonylurea-induced hypoglycaemia: A GoDARTS Study. Diabetes Obes Metab. 2018 Jan;20(1):211-214. doi: 10.1111/dom.13046. Epub 2017 Aug 25. PMID 28656666
- [Background] Wedemeyer RS, Blume H. Pharmacokinetic drug interaction profiles of proton pump inhibitors: an update. Drug Saf. 2014 Apr;37(4):201-11. doi: 10.1007/s40264-014-0144-0. PMID 24550106
- [Background] Semiz S, Dujic T, Ostanek B, Prnjavorac B, Bego T, Malenica M, Marc J, Causevic A. Analysis of CYP2C9*2, CYP2C19*2, and CYP2D6*4 polymorphisms in patients with type 2 diabetes mellitus. Bosn J Basic Med Sci. 2010 Nov;10(4):287-91. doi: 10.17305/bjbms.2010.2662. PMID 21108610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 37 volunteers were recruited in the period between March 4th, 2019 and May 29th, 2019. On May 30th, 2019, volunteers were screened for CYP2C19 genotype status at the General Hospital in Sarajevo, B&H.
Pre-assignment Details: From 23 individuals, CYP2C19 EM/UM metabolisers, 16 were available for further health status assessment. One participant did not meet inclusion criteria and a total of 15 volunteers were randomised.
Period: First Period
Arm/Group | Omeprazole, Then Placebo | Placebo, Then Omeprazole
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Wash-out (10 Days)
Arm/Group | Omeprazole, Then Placebo | Placebo, Then Omeprazole
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0
Period: Second Period
Arm/Group | Omeprazole, Then Placebo | Placebo, Then Omeprazole
Started | 7 | 8
Completed | 7 | 7
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omeprazole, Then Placebo | Placebo, Then Omeprazole | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (3.3) | 21.9 (2.2) | 22.3 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 8 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bosnia and Herzegovina | 7 | 8 | 15
Weight [Mean (Standard Deviation); unit: kilograms] | 82.2 (12.5) | 75.7 (10.8) | 78.7 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Gliclazide AUC
Description: Area under the concentration-time curve (AUC) up to the last concentration measured
Time Frame: 24 hours
Population: A total of 14 participants who completed both study periods were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: μgh/mL
Groups:
- Gliclazide + Omeprazole: Participants received 20 mg of omeprazole alone for 4 days, and concomitantly with single dose of gliclazide on day 5.
- Gliclazide + Placebo: Participants received placebo alone for 4 days, and concomitantly with single dose of gliclazide on day 5.
Arm/Group | Gliclazide + Omeprazole | Gliclazide + Placebo
Number analyzed (Participants) | 14 | 14
μgh/mL | 3.73 [2.81 to 4.93] | 3.29 [2.65 to 4.09]
Statistical Analysis 1: Comparison: Gliclazide + Omeprazole vs Gliclazide + Placebo; The main evaluated outcome was systemic exposure to gliclazide, expressed as AUC(0-t). The geometric mean was calculated for gliclazide AUC(0-24). The ratio of the geometric means with 90% CIs was assessed by linear mixed models between the two treatment assignments: gliclazide and omeprazole co-administration to that of gliclazide and placebo. The obtained 90% CI was compared with the equivalence 0.8-1.25 range; Test type: Equivalence — Sample size calculation was performed using SAS Proc Power procedure for equivalence test in 2x2 crossover design. For an equivalence range of 80-125%, the within-subject coefficient of variation for the AUC values for gliclazide of 7.8% based on previous PK studies, and expected test/reference geometric mean ratios between 87-115%, 14 volunteers (7 individuals per sequence) are required to show the lack of interaction with 85% power; Geometric least square mean ratio = 1.13, 90% CI 2-sided [0.86 to 1.48] — The TOST (two one-sided test) test of equivalence showed that the geometric mean ratio and 90% CI for gliclazide AUC(0-24) between omeprazole and placebo phase was 1.13 (0.86-1.48), with upper confidence limit above the usual 1.25 boundary

2. Secondary Outcome: Glucose
Description: Change in glucose concentration - incremental area under the glucose concentration-time curve from 0 to 12 h
Time Frame: 12 hours
Population: A total of 14 participants who completed both study periods were included in the analysis.
Measure: Mean (Standard Deviation); unit: mmol x h/L
Arm/Group | Gliclazide + Omeprazole | Gliclazide + Placebo
Number analyzed (Participants) | 14 | 14
mmol x h/L | 4.6 (4.3) | 4.0 (3.0)
Statistical Analysis 1: Comparison: Gliclazide + Omeprazole vs Gliclazide + Placebo; Test type: Superiority; p = 0.636, t-test, 2 sided

3. Secondary Outcome: Insulin
Description: Change in insulin concentration - incremental area under the insulin concentration-time curve from 0 to 12 h
Time Frame: 12 hours
Population: A total of 14 participants who completed both study periods were included in the analysis.
Measure: Mean (Standard Deviation); unit: mIU x h/L
Arm/Group | Gliclazide + Omeprazole | Gliclazide + Placebo
Number analyzed (Participants) | 14 | 14
mIU x h/L | 231.6 (93.8) | 265.9 (78.2)
Statistical Analysis 1: Comparison: Gliclazide + Omeprazole vs Gliclazide + Placebo; Test type: Superiority; p = 0.055, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Five days for each intervention.
Arm/Group | Gliclazide + Omeprazole | Gliclazide + Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
Participants received half of the 80 mg gliclazide tablet registered as an immediate-release formulation in Bosnia and Herzegovina (Diprian®, Hemofarm d.o.o. Banja Luka, B&H). However, the concentration-time profiles showed modified-release pattern and incomplete elimination within 24h; thus Cmax, tmax, t1/2, and AUC0-∞ could not be determined. The obtained PK profiles were used at the end for validation of physiologically based pharmacokinetic simulation of omeprazole-gliclazide interaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/48/NCT04198948/Prot_SAP_000.pdf